CLINICAL TRIAL: NCT02152410
Title: Comparison of Two Antalgic Strategies: Acupuncture Versus Intravenous Morphine in the Management of Acute Pain in Emergency Departement. A Randomized Trial of Efficacy and Safety
Brief Title: Acupuncture Versus IV Morphine in the Treatment of Acute Pain in ED
Acronym: AcuMoPE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Monastir (Other)
Collaborators: Emergency NGO Onlus (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 48003/12
Record Dates: First submitted 2013-09-11; First posted 2014-06-02 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Renal Colic
Keywords: acupuncture; renal colic
MeSH Terms: conditions — Renal Colic | interventions — Acupuncture Therapy; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acupuncture group (Experimental): The patient receives acupuncture session lasts between 20 to 30 minutes. Acupuncture will be applied according to the standards for reporting interventions in clinical trials of acupuncture (STRICTA).
  Interventions: Device: acupuncture
- Morphine group (Active Comparator): Each patient must receive a bolus of 5 mg of morphine (5 cc) and 2 mg (2cc) every 10 minutes if no improvement (VAS> 30).
  Interventions: Drug: Morphine

INTERVENTIONS:
Device: acupuncture — Acupuncture will be applied according to the standards for reporting interventions in clinical trials of acupuncture (STRICTA)
  Arms: acupuncture group
Drug: Morphine — bolus of 5 mg of morphine (5 cc) and 2 mg (2cc) every 10 minutes if no improvement of VAS (VAS> 30).
  Arms: Morphine group

SUMMARY:
Renal colics are a common cause af acute intense pain in medical emergency settings requiring often the use of high level antalgics (opioid) to relief the patient.

In the other hand, Acupuncture is well known widely for its therapeutic characteristics, especially in relieving pain.

the aim of these study is to compare this two pain relieving techniques in patients consulting the emergency departement (ED) for acute onset renal colics.

DETAILED DESCRIPTION:
acute onset pain is a frequent cause for consulting the ED (2/3 of patients). renal colics are a common cause for severe acute onset pain, we think approximatively 20% of patients consulting the ED for severe (VAS > 70) acute onset pain have renal colics (RC).

the guidelines for the treatment of severe RC recommend the association of two drugs: a nonsteroidal anti-inflammatory agent (NSAI) typically the Ketoprofen and an antalgic typically opioid (Morphine).

but this one face many critics regarding its safety and tolerance, that's why we investigated other pain relief strategies such as acupuncture.

acupuncture is one of the five branches of the traditional chinese medicine, it has proven its efficacity and safety in many conditions and in RC.

the aim of these study is to assess the feasibility, the safety, and the tolerance of an acupuncture pain-relief strategy compared to the conventional one (intravenous opioids) in the treatment of severe acute onset RC in emergency departement settings.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years

  * has a renal colic
  * VAS over 70
  * has not got another analgesic drug before coming to emergency departement

Exclusion Criteria:

* age under 18 years

  * has not renal colic
  * VAS under 70
  * has got another analgesic treatment before coming to emergency departement
  * fever (T° > 38.5°c)
  * cutaneous infection in the punction sites
  * anuric patient
  * contre indication of morphine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
pain relief by VAS | at baseline, 10, 20, 30, 45 and 60 minutes
  the primary outcome is to assess the efficacity of acupuncture versus IV morphine expressed in VAS reduction during treatment.
  if there is a reduction of more than 50% of the baseline VAS, than the treatment is considered efficient.

SECONDARY OUTCOMES:
side effects | during the 60 minutes of the treatment
  during the 60 minutes of the treatment, we checked the patient for side effects:
  * for morphine: rush, nausea, vomiting, dizziness, dyspnea...
  * for acupuncture: needle fracture, needle retention, muscular contractions... if there are no major side effects noted (vomiting, severe dizziness, allergic reaction, needle fracture) the treatment is considered safe.
number of patients completing the treatment | at baseline
  we calculated the number of patients that accepted the acupuncture treatment versus patient with conventional treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Samir, Professor, Principal Investigator — University hospital of Monastir
Locations (2):
- Tunisia (2):
  - Fattouma Bourguiba University Hospital, Monastir, Monastir Governorate
  - university of Monastir, Monastir, Non-US/Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Lee YH, Lee WC, Chen MT, Huang JK, Chung C, Chang LS. Acupuncture in the treatment of renal colic. J Urol. 1992 Jan;147(1):16-8. doi: 10.1016/s0022-5347(17)37121-5. PMID 1729516
- See also: Acupuncture has a good analgesic effect with a low incidence of adverse reactions. — http://www.ncbi.nlm.nih.gov/pubmed/23213979